CLINICAL TRIAL: NCT06472037
Title: A Prospective, Single-arm, Phase II Study Assessing the Efficacy of Gemcitabine, Nab-paclitaxel, and Cadonilimab With Sequential Short-course Radiotherapy in Locally Advanced Pancreatic Ductal Adenocarcinoma Patients.
Brief Title: AG Combined With Cadonilimab Sequential Short-course Radiotherapy in the Treatment of Locally aPDAC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK104-IIT-C-N1-0122
Record Dates: First submitted 2024-06-18; First posted 2024-06-24 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-06

CONDITIONS: Locally Advanced Pancreatic Ductal Adenocarcinoma
MeSH Terms: interventions — Gemcitabine; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gemcitabine and Nab-paclitaxel combined with Cadonilimab and Sequential Short-course Radiotherapy (Experimental): Cadonilimab 10mg/kg Q3W；Gemcitabine 1000mg/m2 Q4W；Nab-paclitaxel 125mg/m2 Q4W； Short-course Radiotherapy
  Interventions: Drug: Cadonilimab; Drug: Gemcitabine; Drug: Nab-Paclitaxel

INTERVENTIONS:
Drug: Cadonilimab — 10mg/kg，IV，D1，Q3W
  Other Names: AK104
Drug: Gemcitabine — 1000mg/m2，IV，D1、D8、D15，Q4W
  Other Names: Gemcitabine injiection
Drug: Nab-Paclitaxel — 125mg/m2，IV，D1、D8、D15，Q4W
  Other Names: Nab-Paclitaxel-Rituximab Complex

SUMMARY:
A prospective, single-arm, exploratory phase II clinical study evaluating the efficacy of Gemcitabine and Nab-palitaxe combined with Cadonilimab sequential short-course radiotherapy in the treatment of patients with locally advanced pancreatic ductal adenocarcinoma.

DETAILED DESCRIPTION:
This trial is a prospective, single-arm, single-center, phase II clinical study aimed at investigating the efficacy and safety of Cadonilimab combined with Gemcitabine and Nab-palitaxe in short-course radiotherapy neoadjuvant treatment for locally advanced pancreatic ductal adenocarcinoma patients. Patients will receive Gemcitabine and Nab-palitaxe combined with Cadonilimab treatment for one cycle, followed by sequential short-course radiotherapy and then Gemcitabine and Nab-palitaxe combined with Cadonilimab treatment. If feasible, radical surgery will be performed to assess efficacy. A total of 8 cycles of chemotherapy will be administered, followed by Cadonilimab maintenance for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for this study must meet all of the following criteria:

1. Obtain written informed consent before implementing any trial-related procedures;
2. Age ≥ 18 years and ≤ 75 years, gender not specified;
3. Pancreatic cancer confirmed by histopathology examination;
4. Locally advanced pancreatic ductal adenocarcinoma and no prior anti-tumor treatment (radiotherapy, chemotherapy, targeted therapy, immunotherapy, etc.) received;
5. At least one measurable lesion on imaging according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1).
6. ECOG score 0-1;
7. Expected survival time >3 months;
8. Adequate organ function, subjects must meet the following laboratory criteria:

1)Absolute neutrophil count (ANC) ≥1.5x10^9/L without the use of granulocyte colony-stimulating factor in the past 14 days.

2)Platelet count ≥100x10^9/L without blood transfusion in the past 14 days. 3)Hemoglobin > 9g/dL without blood transfusion or use of erythropoietin in the past 14 days; 4)Total bilirubin ≤ 1.5 times the upper limit of normal (ULN); 5)Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 times ULN; 6)Serum creatinine ≤ 1.5 times ULN and creatinine clearance (calculated using the Cockcroft-Gault formula) ≥ 60ml/min; 7)Good coagulation function, defined as international normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 times ULN; 8)Normal thyroid function is defined as thyroid-stimulating hormone (TSH) within the normal range. If the baseline TSH is outside the normal range, subjects with total T3 (or FT3) and FT4 within the normal range may also be included in the study.

9.For female subjects of childbearing potential, a urine or serum pregnancy test should be performed within 3 days before receiving the first dose of the study drug (Day 1 of Cycle 1) and the result should be negative. If the urine pregnancy test result cannot be confirmed as negative, a blood pregnancy test is required. Non-childbearing potential female subjects are defined as postmenopausal for at least 1 year, or having undergone surgical sterilization or hysterectomy.

10.All subjects, male or female, were required to use contraception with an annual failure rate of less than 1% during the entire treatment period up to 120 days after the last dose of study drug (or 180 days after the last dose of chemotherapeutic drug) if there was a risk of pregnancy.

Exclusion Criteria:

1. Malignant diseases other than pancreatic cancer diagnosed within 5 years before the first administration (excluding radical basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and/or carcinoma in situ after radical resection);
2. Is currently participating in an interventional clinical study or has received other study medication or used the study device within 4 weeks prior to the first dose;
3. Prior therapy with anti-PD-1, anti-PD-L1, or anti-PD-L2 drugs or drugs directed against another stimulatory or synergistic T cell receptor suppressor (e.g., CTLA-4, OX-40, CD137);
4. Systemic treatment of Chinese patent medicines with anti-tumor indications or immunomodulatory drugs (including thymosin, interferon and interleukin, except for local use to control ascites) within 2 weeks before the first administration;
5. Active autoimmune disease requiring systemic therapy (e.g., disease-modifying drugs, glucocorticoids, or immunosuppressants) within 2 years prior to the first dose. Replacement therapy (e.g., thyroxine, insulin, or physiologic glucocorticoids for adrenal or pituitary insufficiency) is not considered systemic therapy;
6. Is receiving systemic glucocorticoid therapy (excluding topical glucocorticoids by nasal, inhaled, or other routes) or any other form of immunosuppressive therapy within 7 days prior to the first dose of the study; Note: The use of physiological doses of glucocorticoids (≤10mg/day of prednisone or equivalent) is allowed;
7. Known allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation;
8. Known allergy to the investigational drug carfilzomib, gemcitabine, or any excipient of albumin-bound paclitaxel;
9. Have not fully recovered from any toxicities and/or complications due to any prior interventions before starting treatment (i.e., ≤ Grade 1 or back to baseline, excluding fatigue or alopecia);
10. Known history of human immunodeficiency virus (HIV) infection (i.e., HIV-1/2 antibody positive);
11. Uncontrolled active hepatitis B (defined as HBsAg positive with detectable HBV-DNA copies above the upper limit of normal for the testing laboratory at the study center);

Note: Subjects with the following criteria can also be included:

1. HBV viral load <1000 copies/ml (200 IU/ml) before the first dose, subjects should receive anti-HBV treatment throughout the study drug treatment period to prevent viral reactivation
2. Subjects with anti-HBc (+), HBsAg (-), anti-HBs (-), and HBV viral load (-) do not need to receive prophylactic anti-HBV treatment, but need close monitoring for viral reactivation 12.Subjects with active HCV infection (HCV antibody positive and HCV-RNA levels above the detection limit); 13.Received live vaccines within 30 days before the first dose (Cycle 1, Day 1); Note: Administration of inactivated influenza vaccine for seasonal flu is allowed within 30 days before the first dose, but intranasal live attenuated influenza vaccine is not allowed.

14.Pregnant or lactating women; 15.Presence of any severe or uncontrolled systemic diseases, such as:

1. Resting electrocardiogram showing significant and symptomatic abnormalities in rhythm, conduction, or morphology, such as complete left bundle branch block, second-degree or higher heart block, ventricular arrhythmias, or atrial fibrillation;
2. Unstable angina, congestive heart failure, chronic heart failure with New York Heart Association (NYHA) class ≥2;
3. Any arterial thrombosis, embolism, or ischemia events such as myocardial infarction, unstable angina, cerebrovascular accident, or transient ischemic attack within 6 months prior to initiation of therapy;
4. Suboptimal blood pressure control (systolic blood pressure >140mmHg, diastolic blood pressure >90mmHg);
5. History of non-infectious pneumonia requiring glucocorticoid therapy within 1 year prior to initial dosing, or current clinical active interstitial lung disease;
6. Active pulmonary tuberculosis;
7. Active or uncontrolled infections requiring systemic therapy.
8. Clinical active diverticulitis, intra-abdominal abscess, gastrointestinal obstruction;
9. Liver diseases such as cirrhosis, decompensated liver disease, acute or chronic active hepatitis;
10. Poorly controlled diabetes (fasting blood glucose (FBG) >10mmol/L);
11. Urinalysis shows urine protein ≥++, and confirmed 24-hour urine protein quantification >1.0g;
12. Presence of mental disorders and inability to cooperate with treatment; 16 There may be potential risks that could interfere with the trial results, hinder the full participation of subjects in the study, such as medical history or evidence of diseases, abnormal treatment or laboratory test values, or other conditions deemed unsuitable for inclusion by the researchers. Researchers may also identify other potential risks that make participation in this study unsuitable.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Clinical benefit rate (CBR, CR+PR+SD) | 1 year
  Clinical benefit rate ( complete response and partial response and stable disease)

SECONDARY OUTCOMES:
ORR | 1 yaear
  overall response rate
PCR | 1 year
  Complete pathological response rate
(EFS)RECIST 1.1 | 1 year
  event free survival
OS | 1 year
  Overall survival .OS is defined as the time from date of neoadjuvant treatment start to the date of death from any cause or to the date of last follow-up if patients are alive. If a patient is alive by the time of final analysis, the patient will be censored at the last follow-up date.
Surgical conversion rate | 1 year
  Surgical conversion rate
(AEs)CTCAE 5.0 | 1 year
  Defined as the proportion of patients with AE, treatment-related AE (TRAE), immune-related AE (irAE), serious adverse event (SAE), assessed by NCI CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Rui Liu, MD, Study Chair — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China